CLINICAL TRIAL: NCT02634177
Title: An 8-Week Prospective Randomized, Controlled, Double-Blind Trial of the Genecept Assay ™ vs. Treatment-as-Usual to Evaluate Efficacy of Assay-Guided Treatment in Adults With Major Depressive Disorder (MDD)
Brief Title: Genecept Assay™ vs. Treatment-as-Usual to Evaluate Efficacy of Assay-Guided Treatment in Adults With MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genomind, LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GNM-PROT MDD-01
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
Keywords: Genotyping; Genecept Assay™
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assay-guided treatment (AGT) (Active Comparator): Assay results will be provided to the treating investigator, who will use the results to guide pharmacotherapy of the subject's MDD treatment.
  Interventions: Genetic: Assay-guided treatment (AGT)
- Treatment-as-usual (TAU) (Placebo Comparator): The treating investigator will treat subjects of the TAU group without the knowledge of the pharmacogenetic testing results.
  Interventions: Other: Treatment-as-usual (TAU)

INTERVENTIONS:
Genetic: Assay-guided treatment (AGT) — The assay provides information to guide pharmacotherapeutic decisions personalized to a patient's genetic profile, to maximize improvement in symptomatology and minimize treatment failure and treatment intolerability.
  Other Names: Genecept Assay™
  Arms: Assay-guided treatment (AGT)
Other: Treatment-as-usual (TAU) — Subjects are treated-as-usual without the aid of the assay.
  Arms: Treatment-as-usual (TAU)

SUMMARY:
In this randomized clinical trial, subjects will be assigned to either an assay-guided treatment condition (AGT) or a treatment-as-usual condition (TAU). All subjects will provide a DNA sample at the Screening Visit for the Genecept Assay ™. In the AGT condition, assay results will be provided to the treating investigator, who will use the results to guide antidepressant pharmacotherapy. In the TAU condition, the investigator will treat the subjects without the knowledge of the pharmacogenetic testing results. Assay results for all subjects will be provided to the investigator once all Week 8 visit procedures have been completed. Raters of the primary endpoint assessment and subjects will remain blinded to treatment assignment.

DETAILED DESCRIPTION:
This study compares efficacy and safety outcomes in Major Depressive Disorder (MDD) adult patients randomized to assay-guided treatment (AGT) or treatment-as-usual (TAU). The treatment duration will be 8-weeks. Subjects will be assessed at visits at Week 2, 4, 6 and 8. Approximately 300 subjects will be randomized 1:1 to the two treatment group (AGT and TAU). This is a multi-center trial, with approximately 25 sites in the US. Randomization will be by IWRS. The treating investigator will be unblinded to treatment assignment (necessarily). Other site staff, sponsor staff (including site monitors) and all others will be blinded to treatment assignment for the duration of the subject's participation in the study. The (blinded) rater for the primary endpoint, the SIGH-D-17 Hamilton Depression Scale, will have no other contact with the subject such as collection of screening data, follow-up assessments, documentation of adverse events, etc. Blinded raters will not discuss subjects with other study staff.

After recruitment for main study is completed, an additional 70 subjects , age 65 years and older will be randomized to the Exploratory Elderly MDD Study. This follow-on sub-study will apply all procedures of the main study to this elderly population subset.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years; Sub-Group Age =/> 65 years
2. Ability to understand and provide informed consent
3. Ability to understand, read and speak English
4. Primary diagnosis of Major Depressive Disorder (without psychosis) based on DSM-5 criteria and MINI 7.0
5. SIGH-D-17 score >18 (i.e., moderate depression) at Screening and Baseline
6. Failure of at least 1 prior adequate trial of standard antidepressant in the current major depressive episode (using ATRQ criteria - i.e., 6 weeks at adequate dose) due to inefficacy, side effects or intolerability
7. Subject is willing to follow study instructions, complete study assessments and likely to complete all required visits

Exclusion Criteria:

1. Severe personality traits (based on DSM-5 criteria) that in the opinion of the investigator may interfere with the participation in the study or the evaluation of efficacy and safety and all diagnosed Personality Disorders
2. Current DSM-5 diagnosis of Neurocognitive Disorders, Schizophrenia Spectrum (lifetime diagnosis) and other Psychotic Disorders, Bipolar and Related disorders (lifetime diagnosis*), Trauma and Stress related Disorders, Obsessive Compulsive Disorder and Related Disorders. Other DSM-5 disorders that in the opinion of the investigator may interfere with the participation in the study or the evaluation of efficacy and safety.
3. DSM-5 diagnosis of Substance Related and Addictive Disorders diagnosed in the last 12 months (other than tobacco and caffeine)
4. History of Suicidal Behavior within 12 months of screening or presence of Active Suicidal Ideation with Intent in the past 12 months (Items 4 or 5) at Screening or Baseline, as determined by the Columbia Suicide Severity Rating Scale (C-SSRS), or subject is considered to be an acute suicide risk in the clinical judgment of the investigator
5. Previous homicidal behavior or acute homicidal risk at Screening or Baseline, in the clinical judgment of the investigator
6. Four (4) or more failed pharmacologic interventions for depression in the current major depressive episode (One of the four failed interventions must meet ATRQ criteria - i.e., 6 weeks at adequate dose).
7. Subjects who are not willing to take psychotropic medications for treatment of MDD.
8. Electroconvulsive therapy (ECT) or transcranial magnetic stimulation therapy (TMS) started within 90 days of screening or planned during the study.
9. Subjects with a vagus nerve or deep brain stimulator are prohibited from the trial.
10. Psychotherapy including cognitive behavioral therapy (CBT), or dialectical behavioral therapy (DBT) started within 90 days of screening or planned during the study.
11. Unstable or active medical condition(s) which in the opinion of the investigator would jeopardize the subject's safety or interfere with participation of the study or confound evaluation of efficacy or safety.
12. Current diagnosis of unstable hypothyroidism.
13. Females who are pregnant, nursing, or planning a pregnancy during the study or believe they may be pregnant at Screening or Baseline.
14. Participation in another investigative trial within 30 days of screening
15. Subject previously treated with the use of a similar psychotropic genetic testing assay.
16. Subject tests positive for illicit drug use on the urine drug screen (UDS) at the screen visit (including Marijuana where legal).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Krause, MD, Study Chair — Genomind CMO
Locations (23):
- United States (23):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Noesis Pharma, Phoenix, Arizona
  - Woodland Research Northwest, Springdale, Arkansas
  - Collaborative Neuroscience Network, Inc. - Garden Grove, Garden Grove, California
  - Pacific Institute of Medical Research, Los Angeles, California
  - Pacific Research Partners, LLC, Oakland, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Collaborative Neuroscience Network, Inc. - Torrance, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Florida Clinical Research Center, LLC - Bradenton, Bradenton, Florida
  - Clinical Neuroscience Solutions Inc. - Jacksonville, Jacksonville, Florida
  - Florida Clinical Research Center, LLC - Maitland, Maitland, Florida
  - Clinical Neuroscience Solutions Inc. - Orlando, Orlando, Florida
  - Chicago Research Center, Inc., Chicago, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Richard H Weisler MD, PA and Associates, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Thomas Jefferson University Mood Disorder Program, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions Inc. - Memphis, Memphis, Tennessee
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - University of Virginia Center for Psychiatric Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 304 Randomized
Period: Overall Study
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Started | 151 | 153
Completed | 140 | 141
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Population: The baseline analysis was completed on the all randomized set as defined in the SAP. All data may not have been available for every endpoint for each patient included in the baseline analysis population. Therefore the number of patients at baseline and the number completed may not match specific endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU) | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.38) | 47.6 (12.03) | 47.7 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 111 | 218
  Male | 44 | 42 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 33 | 38 | 71
  White | 111 | 110 | 221
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 151 | 153 | 304
Body Weight (kg) at Screening [Mean (Standard Deviation); unit: kg] | 88.59 (22.338) | 89.28 (24.787) | 88.93 (23.566)
Height at Screening [Mean (Standard Deviation); unit: cm] | 168.3 (10.64) | 168.0 (9.41) | 168.1 (10.03)
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 31.27 (7.491) | 31.62 (8.443) | 31.45 (7.973)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in SIGH-D-17 Score at 8 Weeks.
Description: SIGH-D-17: 17-item rater-administered Structured Interview Guide of the Hamilton Depression Rating Scale
  Scoring is based on the 17-item scale and scores range from 0 minimum to 52 maximum. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale.
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 138 | 140
units on a scale | -9.70 (6.411) | -10.16 (6.689)

2. Secondary Outcome: Mean Change From Baseline in QIDS-SR16 Score at 8 Weeks.
Description: QIDS-SR16: 16-item Quick Inventory of Depressive Symptomatology Self-Report
  QIDS-SR16 ranges from a score of 0 minimum to 27 maximum. In terms of severity of depression, Scores of 0 to 5 reflect "none", scores of 6 to 15 reflect "mild", scores of 7-20 reflect "moderate and scores of 21 to 27 reflect "severe" depression.
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 138 | 141
units on a scale | -6.04 (5.407) | -6.45 (5.135)

3. Secondary Outcome: Percentage of Treatment Responders at Week 8 Based on ≥ 50% Reduction of SIGH-D-17 Score From Baseline.
Description: SIGH-D-17: 17-item rater-administered Structured Interview Guide of the Hamilton Depression Rating Scale
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 138 | 140
Participants | 58 | 72

4. Secondary Outcome: Percentage of Treatment Responders at Week 8 Based on ≥ 50% Reduction of QIDS-SR16 Score From Baseline.
Description: as for outcome 2
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 140 | 141
Participants | 57 | 65

5. Secondary Outcome: Percentage of Treatment Responders at Week 8 Based on ≤ 3 Score on the CGI-I.
Description: CGI-I: Clinical Global Impression Improvement scale; a clinician-rated scale that measures the improvement or worsening of a patient's symptoms
  The CGI-I is rated on a 7-point scale, with the improvement in severity of illness scale using a range of responses from 1 (Very much improved) through to 7 (Very much worse).
  A score of 0 indicates Patient was not able to be assessed
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 140 | 141
Participants | 128 | 118

6. Secondary Outcome: Percentage of Remitters at Week 8 Based on ≤ 7 Score on the SIGH-D-17.
Description: as for outcome 1
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 138 | 140
Participants | 35 | 46

7. Secondary Outcome: Percentage of Remitters at Week 8 Based on ≤ 5 Score on the QIDS-SR16.
Description: as for outcome 2
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 140 | 141
Participants | 43 | 47

8. Secondary Outcome: Safety Outcomes Based on Frequency, Intensity and Burden of Side Effects Rating (FIBSER).
Description: A 3-question patient-rated scale for assessing frequency, intensity, and burden of medication side effects for patients receiving treatment for depression.
  The Frequency, Intensity, and Burden of Side Effects-Rating (FIBSER) questionnaire uses 3 questions with a 6-point Likert measurement scale.
  A score of 0-2 on question 3 (burden of side effects) represents an acceptable low side-effect burden usually requiring no treatment adjustment. A score of 3 or 4 indicates moderate side-effect burden that should be evaluated further (eg, timing related to dose change, patient concerns, etc), and an adjustment such as a dose decrease considered. A score of 5 or 6 indicates a high burden warranting a change such as dose decrease, switching, or direct treatment of the side effect(s).
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 124 | 127
units on a scale | -.02 (1.55) | -.02 (1.55)

9. Secondary Outcome: Safety Outcomes Based on Frequency and Severity of Reported Adverse Events.
Description: Untoward medical occurrence in a subject administered a pharmaceutical product which does not necessarily have to have a causal relationship with treatment.
  As based on FIBSER
  The Frequency, Intensity, and Burden of Side Effects-Rating (FIBSER) questionnaire uses 3 questions with a 6-point Likert measurement scale.
  A score of 0-2 on question 3 (burden of side effects) represents an acceptable low side-effect burden usually requiring no treatment adjustment. A score of 3 or 4 indicates moderate side-effect burden that should be evaluated further (eg, timing related to dose change, patient concerns, etc), and an adjustment such as a dose decrease considered. A score of 5 or 6 indicates a high burden warranting a change such as dose decrease, switching, or direct treatment of the side effect(s). Scores refer to intensity, frequency and interference.
Time Frame: Screening to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 124 | 127
score on a scale
  Frequency of the side effects for the past week | -0.1 (2.18) | -0.2 (2.18)
  Intensity of the side effects over the last week | 0.0 (1.86) | 0.0 (1.9)
  Interference of day-to-day functions over the last | -0.2 (1.55) | -0.2 (1.59)

ADVERSE EVENTS:
Time Frame: AEs were collected at all study visits screening to Week 8
Description: Adverse Events were based on the "Safety Analysis Set: All randomized subjects who complete the (post-randomization) baseline appointment with the treating investigator, i.e., start AGT or TAU treatment
Arm/Group | Assay-guided Treatment (AGT) | Treatment-as-usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/153
Serious Adverse Events (participants affected / at risk) | 6/150 | 3/153
Other Adverse Events (participants affected / at risk) | 107/150 | 111/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assay-guided Treatment (AGT) (N=150) | Treatment-as-usual (TAU) (N=153)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assay-guided Treatment (AGT) (N=150) | Treatment-as-usual (TAU) (N=153)
Headache (Nervous system disorders) | 22 (22) | 15 (15)
Dizziness (Nervous system disorders) | 13 (13) | 19 (19)
Somnolence (Nervous system disorders) | 5 (5) | 10 (10)
Sedation (Nervous system disorders) | 7 (7) | 4 (4)
Coordination abnormal (Nervous system disorders) | 2 (2) | 6 (6)
Tremor (Nervous system disorders) | 2 (2) | 6 (6)
Dizziness postural (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2)
Hypersomnia (Nervous system disorders) | 1 (1) | 2 (2)
Tension headache (Nervous system disorders) | 3 (3) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Narcolepsy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 22 (22) | 15 (15)
Nausea (Gastrointestinal disorders) | 15 (15) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 14 (14)
Constipation (Gastrointestinal disorders) | 13 (13) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feces soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 9 (9)
Anxiety (Psychiatric disorders) | 9 (9) | 7 (7)
Irritability (Psychiatric disorders) | 6 (6) | 10 (10)
Libido decreased (Psychiatric disorders) | 3 (3) | 9 (9)
Restlessness (Psychiatric disorders) | 4 (4) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 4 (4)
Bruxism (Psychiatric disorders) | 3 (3) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 1 (1)
Anorgasmia (Psychiatric disorders) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 1 (1) | 2 (2)
Middle insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Orgasm abnormal (Psychiatric disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Derealisation (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 (11) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Pruritus (Infections and infestations) | 3 (3) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 4 (4)
Chest pain (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Edema peripheral (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 5 (5) | 4 (4)
Dysuria (Renal and urinary disorders) | 5 (5) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Micturition frequency decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 5 (5) | 4 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 7 (7)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Cardiac disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nocturnal emission (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT02634177/SAP_000.pdf
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02634177/Prot_001.pdf